CLINICAL TRIAL: NCT00618514
Title: Comparative Evaluation of the FDA-Cleared Bright Tip Laser Fiber Versus Commercially Available Bare Laser Fiber (the Control) in the Treatment of Reflux in the Greater Saphenous Vein (GSV) Using Endovenous Laser Therapy
Brief Title: The BRILLIANT Study
Acronym: BRILLIANT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Vascular Solutions LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0407
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2013-06

CONDITIONS: Varicose Veins
Keywords: Varicose Veins; Laser Ablation; Laser Wire Fibers
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Bright Tip Laser Fiber - FDA-cleared study device
  Interventions: Device: Bright Tip Laser Fiber
- 2 (Active Comparator): Standard bare tip Laser Fiber - Any commercially available laser device (the control)
  Interventions: Device: Bare Tip Laser Fiber

INTERVENTIONS:
Device: Bright Tip Laser Fiber — Endovenous laser ablation treatment for varicose veins in a section of the Greater Saphenous Vein (GSV) using a laser fiber with a fitted ceramic tip on the end. Treatment performed on one leg.
  Arms: 1
Device: Bare Tip Laser Fiber — Endovenous laser ablation treatment for varicose veins in a section of the Greater Saphenous Vein (GSV) using a laser fiber readily available on the market with a bare tip on the end. Treatment performed on one leg.
  Arms: 2

SUMMARY:
This trial was designed as a prospective, multi-center, randomized clinical trial of the FDA-cleared Vari-Lase Bright Tip Fiber compared to commercially available standard bare-tip laser fiber (control) to demonstrate the safety and effectiveness of laser ablation for the treatment of varicose veins associated with reflux within the great saphenous vein (GSV) and to provide additional data concerning patient satisfaction. Within this evaluation, subject limbs were randomized to one of two (2) treatment groups utilizing a 1:1 randomization ratio. If a subject required treatment of only one limb, that limb was randomized to a treatment group. If a subject required treatment of two limbs, the first limb was randomly assigned treatment and the second limb was assigned the other treatment (the opposite treatment of the other limb). The data was analyzed by treated limb (versus treated subject).All study data were analyzed under the principles of intent-to-treat, in which data are analyzed according to the assigned randomized group regardless of the treatment actually delivered. Subjects were followed at one week, one month, and six months.

DETAILED DESCRIPTION:
This trial was designed as a prospective, multi-center, randomized clinical trial of the FDA-cleared Vari-Lase Bright Tip Fiber compared to commercially available standard bare-tip laser fiber (control) to demonstrate the safety and effectiveness of laser ablation for the treatment of varicose veins associated with reflux within the great saphenous vein (GSV) and to provide additional data concerning patient satisfaction. Subjects were pre-screened utilizing standard of care data (including documented evidence of reflux within the GSV) for the specified inclusion/exclusion criteria to ensure that they were eligible for treatment in the investigation. Prior to laser treatment and after signing an informed consent form, study eligibility assessments were completed including physical assessment of target limb(s), duplex ultrasound of GSV segment(s) targeted for treatment, symptom assessment, medical history, and digital photos of targeted limbs. Upon enrollment, targeted limbs were randomized at a 1:1 ratio to receive the Vari-lase Bright Tip Fiber or the control treatment. If the subject required treatment of two limbs, the first limb was randomized and the second limb was assigned the other treatment (the opposite treatment of the other limb). Immediately post procedure, subjects were assessed for adverse events and a physical assessment of the treated limb(s) was performed. Subjects were also asked to complete a subject pain and satisfaction questionnaire. Subjects were followed at one week, one month, and six months. Follow-up included a physical assessment of treated limb(s), symptom assessment, adverse event assessment, and completion of a subject pain and satisfaction questionnaire. Additionally, a duplex ultrasound assessment was conducted at one week and six months and digital photos were taken of the treated vein segment(s) at one week and one month. The data was analyzed by treated limb (versus treated subject). All study data were analyzed under the principles of intent-to-treat, in which data are analyzed according to the assigned randomized group regardless of the treatment actually delivered.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older
2. Subjects with primary varicose veins resultant of GSV reflux documented on duplex ultrasound
3. Subjects that will be undergoing endovenous laser ablation treatment of varicose veins
4. Subjects treatment includes the Greater Saphenous Vein
5. If bilateral, subject is willing and able to undergo treatment of both legs within two weeks.
6. Subjects who are willing and able to comply with the requirements of the study protocol
7. Subjects who are willing and able to provide informed consent

Exclusion Criteria:

1. Subjects with severe peripheral vascular disease (PVD) as evidenced by an ankle-brachial index of < 0.5
2. Subjects who are unable to ambulate at baseline
3. Subjects with thrombosis in the vein segment(s) to be treated
4. Subjects that have had prior vein treatment
5. Subjects who are known or suspected to be pregnant or lactating
6. Subjects that are concurrently participating in an investigational study that may confound the treatment or outcomes of the present study
7. Subjects with an active or systemic infection
8. Anatomic variants- duplication of the GSV, presence of incompetent accessory veins of the GSV
9. Subjects who are scheduled to have a bilateral treatment, where one limb is to be enrolled in this study and the second limb that is not treated as part of this study, is treated within two months of the procedure for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Worthington-Kirsch, MD, Principal Investigator — Image Guided Surgery Associates
Locations (7):
- United States (7):
  - Southeast Vein and Laser, Dothan, Alabama
  - Morrision Vein Institute, Scottsdale, Arizona
  - HealthwoRx, Hollywood, Florida
  - Mackay Center for Vein Treatment and Laser Therapy, Palm Harbor, Florida
  - Comprehensive Wound Care, Kinston, North Carolina
  - Pottstown Memorial Hospital, Pottstown, Pennsylvania
  - The Vein Center of Virginia, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who had a planned endovenous laser ablation treatment for varicose veins that included treatment of the Greater Saphenous Vein (GSV) were recruited from medical clinics.
Pre-assignment Details: 93 subjects enrolled, 3 subjects were not randomized because they withdrew consent prior to receiving study procedure; 90 subjects randomized and 110 limbs were assigned treatment.
Groups:
- Bright Tip Laser Fiber: Investigational Device: The laser fiber is positioned at least two cm distal to the saphenofemoral junction. Laser energy is delivered through the 810 nm diode laser set at 10-14 watts. Subjects in this category had only one limb treated with the Bright tip laser fiber.
- Standard Bare Tip Laser Fiber: Control Device: The laser fiber is positioned at least two cm distal to the saphenofemoral junction. Laser energy is delivered through the 810 nm diode laser set at 10-14 watts. Subjects in this arm had only one limb treated with the bare tip laser fiber (control).
- Bright Tip Laser & Bare Tip Laser: Subjects that received testament of both limbs using the investigational device (Bright Tip laser) and the control (bare tip laser)
Period: Overall Study
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber | Bright Tip Laser & Bare Tip Laser
Started | 36 | 38 | 16
Completed | 25 | 26 | 12
Not Completed | 11 | 12 | 4
Not completed — Lost to Follow-up | 11 | 12 | 4

BASELINE CHARACTERISTICS:
Population: Reporting per limb treated (versus per subject)
Groups:
- Bright Tip Laser Fiber: Investigational Device: The laser fiber is positioned at least two cm distal to the saphenofemoral junction. Laser energy is delivered through the 810 nm diode laser set at 10-14 watts.
- Standard Bare Tip Laser Fiber: Control Device: The laser fiber is positioned at least two cm distal to the saphenofemoral junction. Laser energy is delivered through the 810 nm diode laser set at 10-14 watts.
- Total: Total of all reporting groups
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (12.7) | 53.8 (14.1) | 54.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 44 | 84
  Male | 15 | 11 | 26
Region of Enrollment [Number; unit: Limbs]
  United States | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Limbs With a Continued Absence of Flow Within the Treated Vein Segment Over 6 Months.
Description: The absence of flow was evaluated in each treated limb and determined by ultrasound (duplex or Doppler) interrogation.
Time Frame: 6 Months
Measure: Number; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber
Number analyzed (Participants) | 38 | 37
Number analyzed (Limbs) | 38 | 37
Limbs | 36 | 36

2. Primary Outcome: Number of Limbs With a Device-related Serious Adverse Event Reported Over 6 Months.
Description: Each treated limb was clinically evaluated for the presence of a device-related serious adverse event.
Time Frame: 6 Months
Measure: Number; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber
Number analyzed (Participants) | 54 | 52
Number analyzed (Limbs) | 54 | 52
Limbs | 0 | 0

3. Secondary Outcome: Percent Change of Subject Symptoms in Treated Limb From Baseline to 6 Months Using Venous Clinical Severity Score (VCSS).
Description: VCSS is a physician's evaluation of 10 pre-determined clinical signs or attributes of venous disease (pain, varicose veins, venous edema, skin pigmentation, inflammation, induration, number of active ulcers, active ulcer duration, active ulcer diameter and compression therapy). Each attribute receives a score from 0-3 (0=absent and 3=severe). The best total overall score is 0 (all ten attributes are absent) and the worse overall score is 30 (all ten attributes are severe). Each treated limb was evaluated and scored at baseline and at 6 months.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage change
Units Other Than Participants: Limbs
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber
Number analyzed (Participants) | 39 | 37
Number analyzed (Limbs) | 39 | 37
percentage change | -64.1 (22.5) | -59.4 (34.8)

4. Secondary Outcome: Percent Change of Subject Symptoms in Treated Limb From Baseline to 6 Months Using Venous Disability Score (VDS).
Description: VDS is a physician's evaluation of a patient's ability to work an eight-hour day with or without a support device (i.e., compressive therapy, limb elevation). The patient is scored on a scale of 0-3 (0=asymptomatic and 3=unable to carry out usual activities (patients activities before the onset of disability due to venous disease) even with compression and/or limb elevation). The score represents the degree of disability caused by the venous disease with the best score being 0 and the worse score being 3. Each treated limb was evaluated and scored at baseline and at 6 months.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage of change
Units Other Than Participants: Limbs
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber
Number analyzed (Participants) | 38 | 35
Number analyzed (Limbs) | 38 | 35
percentage of change | -39.3 (25.5) | -47.1 (19.2)

5. Secondary Outcome: Percent Change of Subject Symptoms in Treated Limb From Post-procedure to 6 Months Using Patient Visual Analog Scale (VAS) Pain Scores.
Description: Each subject completed a questionnaire to rate his/her pain. The scale is from 0-10 (0=no pain and 10=worst pain imaginable). Each treated limb was scored by the patient post-procedure and at 6 months to determine the improvement after treatment at the 6-month time point.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage of change
Units Other Than Participants: Limbs
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber
Number analyzed (Participants) | 40 | 36
Number analyzed (Limbs) | 40 | 36
percentage of change | -35.8 (54.8) | -44.9 (44.8)

6. Secondary Outcome: Percentage of Subjects Reporting an Excellent Satisfaction Score at 6 Months.
Description: Each subject completed a questionnaire to rate their satisfaction with the laser treatment. The score was reported as excellent, good, fair or poor. The best score of excellent was defined as "I am very satisfied with the laser treatment" and the worse score of poor was defined as "I am not satisfied with the laser treatment." Each treated limb was scored by the patient at 6 months to determine the percent satisfaction at the 6-month time point.
Time Frame: 6 months
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Patients
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber
Number analyzed (Participants) | 40 | 37
Number analyzed (Patients) | 40 | 37
Percentage of participants
  Excellent Patient Satisfaction Score | 72.5 | 64.9
  Good Patient Satisfaction Score | 15.0 | 29.7
  Fair Patient Satisfaction Score | 7.5 | 2.7
  Poor Patient Satisfaction Score | 5.0 | 2.7

7. Secondary Outcome: Number of Limbs With a Device-related Non-serious Adverse Event Reported Over 6 Months.
Description: Each treated limb was clinically evaluated for the presence of a device-related non-serious adverse event.
Time Frame: 6 Months
Measure: Number; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber
Number analyzed (Participants) | 54 | 52
Number analyzed (Limbs) | 54 | 52
Limbs | 2 | 1

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Subjects were assessed for adverse events at 1-week, 1-month and 6-month follow-up office visits.
Arm/Group | Bright Tip Laser Fiber | Standard Bare Tip Laser Fiber
Serious Adverse Events (participants affected / at risk) | 0/54 | 1/52
Other Adverse Events (participants affected / at risk) | 3/54 | 2/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bright Tip Laser Fiber (N=54) | Standard Bare Tip Laser Fiber (N=52)
Death (General disorders) | 0 | 1 — Unknown cause of death; this death was reported at 12 months (6 months after the last study required visit)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bright Tip Laser Fiber (N=54) | Standard Bare Tip Laser Fiber (N=52)
Recanalization (Vascular disorders) | 3 | 2

LIMITATIONS AND CAVEATS:
Due to budgetary constraints, enrollment in the BRILLIANT trial was ended after 90 subjects (110 limbs) were enrolled in the study. This study had an insufficient sample size to perform the planned formal statistical hypothesis testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less